CLINICAL TRIAL: NCT06513832
Title: Asthma Navigator Intervention to Improve Health Equity in Children
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Georgia Clinical & Translational Science Alliance (CTSA) (Unknown)
Responsible Party: Principal Investigator, Anne M Fitzpatrick, Assistant Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: STUDY00007482
Record Dates: First submitted 2024-07-15; First posted 2024-07-22 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Asthma in Children
Keywords: Asthma self-management; Asthma in Children

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The study team and participants will not be blinded but statistical analyses will be performed in a blinded fashion using allocations of "Intervention A" and "Intervention B." Randomization will be implemented 2:1, in blocks of 6, via a computer algorithm to minimize unintentional imbalances between groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The Asthma Navigator (Experimental): The Children's electronic medical record (EMR) of each child will be screened weekly for up to 52 weeks. When an asthma exacerbation prompting unscheduled healthcare utilization is noted (primary outcome), or at the end of 52 weeks, participant involvement in the study will end.
  Interventions: Behavioral: The asthma navigator
- Standard of Care (No Intervention): This arm will not have access to the Asthma Navigator.
  The Children's EMR of each child will be screened weekly for up to 52 weeks. When an asthma exacerbation prompting unscheduled healthcare utilization is noted (primary outcome), or at the end of 52 weeks, participant involvement in the study will end.

INTERVENTIONS:
Behavioral: The asthma navigator — The asthma navigator is a Registered Respiratory Therapist and Certified Asthma Educator who will review the care plan at discharge and provide asthma education; assist with follow-up clinic appointment scheduling, medication access, and transportation; and daily as-needed telephone support.
  Arms: The Asthma Navigator

SUMMARY:
The goal of this study is to improve health equity in children aged 5-16.9 years admitted to the PICU for asthma. The objectives are:

* To identify the factors related to differential experiences of asthma self-management
* To pilot the effectiveness of an individualized asthma navigator intervention at PICU discharge.

DETAILED DESCRIPTION:
Despite available asthma treatments, nearly 50% of children with asthma experience exacerbations annually, with disadvantaged children, particularly Black and Hispanic, being the most affected. These disparities are largely due to social determinants of health (SDOH), including socioeconomics and family hardship, which explain over 80% of the racial disparities in asthma outcomes. Children in lower opportunity neighborhoods face additional challenges like poor housing and limited green spaces, increasing exposure to pollutants and allergens.

At Children's Healthcare of Atlanta's Pediatric ICU (PICU), 85% of asthma admissions come from low-opportunity areas, with 36.7% having another exacerbation within a year. Significant barriers to better outcomes include limited provider understanding of SDOH and challenges in asthma self-management. Effective asthma self-management, supported by medical providers, is crucial for improving health outcomes in these disadvantaged children.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to the PICU for asthma

Exclusion Criteria:

* Cystic fibrosis
* Immune deficiency
* Prematurity <35 weeks
* Gestation and congenital airway deformities
* Non-English speaker

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 75 (Estimated)
Dates: Start 2025-01-17 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Future unscheduled healthcare utilization for asthma exacerbation | Baseline, end of study (average of 52 weeks)
  The occurrence of unscheduled healthcare utilization and the date and time of occurrence will be assessed through weekly screenings of each child's EMR at Children's (Epic system).

OTHER OUTCOMES:
Hospitalization occurrence | Baseline, end of study (average of 52 weeks)
  Number of hospitalizations would be measured.
Clinic follow-up | Baseline, end of study (average of 52 weeks)
  Number of clinic follow ups would be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Anne Fitzpatrick, PhD, APRN, Principal Investigator — Emory University
Locations (1):
- Children's Healthcare of Atlanta, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
All subject-level clinical data at enrollment will be preserved and shared during study completion on 7/31/26. Shared data will be deidentified and original data maintained at the Principal Investigator's institution. Recruitment progress and final study results will be documented at clinicaltrials.gov. Protocols, informed consent forms to participate in the trial and the data dictionary will be shared with the data. Data will be shared with qualified investigators with an appropriate research and approved data use agreement (DUA). Data will be accessed by restricted download once approved.
Supporting Information: Study Protocol, ICF
Time Frame: At the time of study completion on August 2026
Access Criteria: Data will be accessed by restricted download once approved.